CLINICAL TRIAL: NCT03730688
Title: Non-invasive Limb Compartment Pressure Measurement
Acronym: FNO-TRAUMA-CPM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Ostrava (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FNO-TRAUMA-CPM; RVO-FNOs/2018 (Other Grant/Funding Number: University Hospital Ostrava)
Record Dates: First submitted 2018-11-02; First posted 2018-11-05 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-12

CONDITIONS: Compartment Syndromes; Polytrauma; Burn Injury
Keywords: compartment syndrome; compartment pressure; polytrauma; burn injury; limb ischemia; fasciotomy
MeSH Terms: conditions — Compartment Syndromes; Multiple Trauma; Burns

STUDY DESIGN:
Intervention Model Description: Compartment pressure will be measured in a single group of patients, using the conventional and the newly developed experimental means of measurement.
Masking Description: No masking will be used in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Conventional and experimental compartment pressure measurement (Experimental): Compartment pressure in the patients in this group will be measured using the conventional Intra-Compartmental Pressure Monitor System (Stryker) and using the newly-developed measuring device.
  Interventions: Device: Conventional compartment pressure measurement; Device: Experimental compartment pressure measurement

INTERVENTIONS:
Device: Conventional compartment pressure measurement — Compartment pressure will be measured using the conventional compartment pressure measurement system.
Device: Experimental compartment pressure measurement — Compartment pressure will be measured using the newly-developed compartment pressure measurement system.

SUMMARY:
Compartment syndrome (CS) is a serious complication of soft-tissue injuries in patients with fractures of the musculoskeletal apparatus. CS is defined as a condition, during which an increased tissue pressure inside an enclosed compartment damages the microcirculation and neuromuscular function of the tissue, and results in ischemization, with a damage of nerve-muscle structures, which lead either to extensive flexion contractures, or myonecroses, with the need to perform an early amputation of the affected limb. In traumatology, compartment syndrome is most frequently observed in a patient with crural fractures, closed as well as open fractures, or in cases of crus laceration.

DETAILED DESCRIPTION:
Compartment syndrome (CS) is a serious complication of soft-tissue injuries in patients with fractures of the musculoskeletal apparatus. CS is defined as a condition, during which an increased tissue pressure inside an enclosed compartment damages the microcirculation and neuromuscular function of the tissue, and results in ischemization, with a damage of nerve-muscle structures, which lead either to extensive flexion contractures, or myonecroses, with the need to perform an early amputation of the affected limb. In traumatology, compartment syndrome is most frequently observed in patients with crural fractures, closed as well as open fractures, or in cases of crus laceration. Diagnostics of the compartment syndrome is very difficult, even today, when numerous emergency osteosyntheses are performed, as it depends not only on the clinical examination of the injured patient but also upon subjective symptoms, which may not be always clearly apparent and objectively quantifiable in a disoriented patient with concussion, or in an unconscious patient. At present, intracompartmental pressure is measured with invasive techniques only (with the insertion of the measurement needle into the compartment space, and administration of saline), or invasively, using piezoelectric probes, similarly to a measurement of pressure in vessels. Both these techniques are invasive, and as such may be associated with complications (infection at the puncture site, increase of intracompartmental pressure with administration of the measuring liquid, or formation of haematoma and bleeding at the probe site).

Physiological values of intracompartmental pressure vary between 5 and 10 mmHg, in case an increase over 20 mmHg is observed, emergency dermatofasciotomy is indicated.

The presented project is aimed at comparing the invasive and non-invasive techniques of compartment syndrome measurement.

The aim of the project is to develop a new non-invasive examination technique of intracompartmental pressure measurement in soft tissues of the injured extremity, with the possibility of its observation and continuous monitoring of the measured values.

Partial aims

1. Invasive measurement of limb intracompartmental pressure.
2. Development of a new examination technique for non-invasive measurement of the compartment syndrome, in cooperation with researchers from the Technical University Ostrava
3. Measurement of compartment syndrome using the new non-invasive examination technique and monitoring of data

Methods First of all, compartmental pressures in the limbs will be performed using the invasive technique. The measurement will be performed also in cases when a fasciotomy was indicated and performed, and the authors will monitor the decrease of compartmental pressure in the course of treatment. Individual measurements will be recorded and statistically analyzed. In the course of measurement, the researchers will work upon the development of a new non-invasive examination technique, which will be intended for non-invasive measurement of compartmental pressure. The research team will also compare both these techniques, and assess the advantages and disadvantages of each of the techniques used.

Statistical data processing Results of measurements of compartmental pressure using individual techniques will be statistically evaluated, depending on the clinical findings at the injured extremity.

ELIGIBILITY:
Inclusion Criteria:

* polytrauma
* monotrauma
* burn injury

Exclusion Criteria:

* age below 15 years of age
* skin infection at the area of measurement
* limb-loss trauma

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
A 30% decrease of complications related to compartment pressure measurement | 37 months
  The number of complications related to compartment pressure measurement will be observed for both interventions, with the target of achieving a 30% decrease.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Novák, MD, Principal Investigator — University Hospital Ostrava
Locations (2):
- Czechia (2):
  - Technical University Ostrava, Ostrava, Moravian-Silesian Region
  - University Hospital Ostrava, Ostrava, Moravian-Silesian Region

IPD SHARING:
Plan to Share IPD: Undecided
The study team have not decided to make individual participant data available to other researchers.

REFERENCES:
- [Background] Beniwal RK, Bansal A. Osteofascial compartment pressure measurement in closed limb injuries - Whitesides' technique revisited. J Clin Orthop Trauma. 2016 Oct-Dec;7(4):225-228. doi: 10.1016/j.jcot.2016.01.001. Epub 2016 Feb 10. PMID 27857494
- [Background] Wiemann JM, Ueno T, Leek BT, Yost WT, Schwartz AK, Hargens AR. Noninvasive measurements of intramuscular pressure using pulsed phase-locked loop ultrasound for detecting compartment syndromes: a preliminary report. J Orthop Trauma. 2006 Jul;20(7):458-63. doi: 10.1097/00005131-200608000-00002. PMID 16891936
- [Background] Dickson KF, Sullivan MJ, Steinberg B, Myers L, Anderson ER 3rd, Harris M. Noninvasive measurement of compartment syndrome. Orthopedics. 2003 Dec;26(12):1215-8. doi: 10.3928/0147-7447-20031201-11. PMID 14690292
- [Background] Lee SH, Padilla M, Lynch JE, Hargens AR. Noninvasive Measurements of Pressure for Detecting Compartment Syndromes. J Orthop Rheumatol. 2013 Dec 21;1(1):5. PMID 25328908